CLINICAL TRIAL: NCT03350243
Title: Coached, Coordinated, Enhanced Neonatal Transition (CCENT): A Multi-centre Mixed-methods Pragmatic Randomized Controlled Trial
Brief Title: Coached, Coordinated, Enhanced Neonatal Transition (CCENT)
Acronym: CCENT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Collaborators: Sunnybrook Health Sciences Centre (Other); Children's Hospital of Eastern Ontario (Other); MOUNT SINAI HOSPITAL (Other); The Ottawa Hospital (Other); Montreal Children's Hospital of the MUHC (Other); Provincial Health Services Authority British Columbia (Other)
Responsible Party: Principal Investigator, Julia Orkin, Staff Physician, Medical Director of the Complex Care Program, The Hospital for Sick Children
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 1000057100
Record Dates: First submitted 2017-11-01; First posted 2017-11-22 (Actual); Last update posted 2023-04-13 (Actual); Status verified 2023-04

CONDITIONS: Prematurity
Keywords: Neonatal Intensive Care Unit; Mindfulness; Care coordination; Anticipatory guidance; Parental support; Neonatal follow-up; Acceptance and Commitment Therapy
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CCENT Intervention group (Experimental): Participants will be assigned a dedicated key worker that will support families through the child's first year, in addition to standard medical care, which involves a primary care provider and/or neonatal follow-up at routine times.
  Interventions: Other: CCENT Intervention
- Control group (No Intervention): Participants will receive the standard medical care at their institution, which involves a primary care provider and/or neonatal follow-up at routine times.

INTERVENTIONS:
Other: CCENT Intervention — 1. Acceptance and Commitment Therapy approach: engaging families through structured individual or group sessions within the NICU and continue this support once discharged.
  2. Care coordination: supporting providers in clear communication when liaising across various levels of care as well as supporting families in system and resource navigation.
  3. Anticipatory guidance: proactive education targeting normal challenges in caring for a child who required intensive care support.
  Arms: CCENT Intervention group

SUMMARY:
This study will evaluate a new neonatal follow-up model that offers additional support and coping resources for parents during their child's NICU admission as well as during their transition home. The Coached, Coordinated, Enhanced Neonatal Transition (CCENT) model involves a key worker who will be the primary support for families during the first year of their child's life. The key worker's role involves 1) parental coaching using an Acceptance and Commitment Therapy approach, 2) coordinating care across various levels of care as well as supporting families in system and resource navigation, and 3) provided proactive education targeting normal challenges in caring for a child who required intensive care support. The goal is to improve the psychosocial support and medical care coordination beyond the neonatal intensive care unit as many of the medical and social concerns do not end at the time of discharge. Primary objective is parent stress at 12 months.

ELIGIBILITY:
Inclusion Criteria (meets at least one of the following criteria):

1. Infant born ≤ 26+6 weeks of gestational age (GA)
2. Infant born between 27-29+6 weeks GA with ≥ 1 of the following risk factors:

   i)≥ Grade III intraventricular hemorrhage with post hemorrhagic hydrocephalus ii)Retinopathy of prematurity requiring intraocular bevacizumab/ anti-vascular endothelial growth factor or laser surgery therapy iii)Requires invasive (e.g., intubated) or non-invasive (e.g., CPAP or BiPAP) at ≥ 34 weeks GA and/or supplemental oxygen at ≥ 37 weeks gestational age iv)Requires surgery for management of necrotizing enterocolitis (NEC)- stage 3
3. Infant with ≥ 2 major congenital anomalies as defined by EUROCAT(13) (e.g., congenital heart disease, spina bifida, cleft palate, etc. Not including minor congenital anomalies, e.g., dysmorphic facies), and length of stay in recruiting institution ≥ 14 days.
4. Infant with hypoxic ischemic encephalopathy (HIE) requiring therapeutic hypothermia and in the recruiting institution for ≥ 14 days.

Exclusion Criteria:

1. Families that do not speak English or French
2. Parent will not be involved with child's care over the entirety of the study period (2 years) (e.g., adoption).
3. Infant will be followed by an out-of-province neonatal follow-up program or lives a significant distance from the neonatal follow up program and therefore not routinely followed by the team.
4. Infant that has previously been discharged home from the NICU/hospital.
5. Decision/high likelihood of decision for act of withdrawal of care by clinical teams/families

Ages: 0 Months to 4 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 275 (Actual)
Dates: Start 2018-01-31 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-10-31 (Actual)

PRIMARY OUTCOMES:
Change in Parental Stress | 12 months
  This outcome will be assessed using the Parenting Stress Index 4th Edition (PSI-4) Short Form questionnaire.

SECONDARY OUTCOMES:
Parental Quality of Life (QoL) | 4 months
  The Health Utilities Index (HUI) questionnaire provides a health-related quality of life (HRQL) score for overall health, which will be used to calculate quality-adjusted life years (QALYs) for a cost-utility analysis.
Parental Quality of Life (QoL) | 12 months
  The Health Utilities Index (HUI) questionnaire provides a health-related quality of life (HRQL) score for overall health, which will be used to calculate quality-adjusted life years (QALYs) for a cost-utility analysis.
Parental Empowerment | 12 months
  This outcome will be assessed using the Family Empowerment Scale (FES), which measures empowerment across three specific domains: 1) family, 2) service system, and 3) community/political.
Child Social and Emotional Development | 12 months
  This outcome will be assessed using the Brief Infant-Toddler Social Emotional Assessment (BITSEA), which is a parent self-report questionnaire that is designed as a screener to identify children (1-3 years old) at risk for or currently experiencing social-emotional and/or behavioural problems.
Parent and Child Interaction | 12 months
  This outcome will be assessed using the Nursing Child Assessment Satellite Training Parent-Child Interaction (NCAST-PCI), which is used assess caregiver and infant behaviour during a structured teaching task.
Maternal Depression | 6 weeks
  This outcome will be assessed using the Edinburgh Postnatal Depression Scale (EPDS), which is a screening tool used to identify those with symptoms associated with postnatal depression in the previous 7 days. Composite score between 0 to 30 will be recorded, with a score of 10 or greater indicating possible depression.
Maternal Depression | 4 months
  This outcome will be assessed using the Edinburgh Postnatal Depression Scale (EPDS), which is a screening tool used to identify those with symptoms associated with postnatal depression in the previous 7 days. Composite score between 0 to 30 will be recorded, with a score of 10 or greater indicating possible depression.
Maternal Depression | 12 months
  This outcome will be assessed using the Edinburgh Postnatal Depression Scale (EPDS), which is a screening tool used to identify those with symptoms associated with postnatal depression in the previous 7 days. Composite score is given between 0 to 30. Possible depression is a score of 10 or greater.
Child Development | 18 months
  The Bayley Scales of Infant and Toddler Development (3rd Edition) will be used to assess neurodevelopment with separate composite scores (mean 100 ± SD 15) for cognition, language, and motor skills.
Healthcare Service Delivery | 12 months
  This outcome will be assessed using the Measure of Processes of Care (MPOC20) questionnaire, which is used to measure the parent's perception of the health services they and their child receive.
Maternal Anxiety | 4 months
  This outcome will be assessed using the State-Trait Anxiety Inventory (STAI) questionnaire, which often used in research as an indicator of caregiver distress.
Maternal Anxiety | 12 months
  This outcome will be assessed using the State-Trait Anxiety Inventory (STAI) questionnaire, which often used in research as an indicator of caregiver distress.
Resource Utilization | 4 months
  The Resource Use Questionnaire (RUQ) will assess family resource use relating to their child's medical needs, services and programs, as well as parent time losses and family out-of-pocket costs.
Resource Utilization | 12 months
  The Resource Use Questionnaire (RUQ) will assess family resource use relating to their child's medical needs, services and programs, as well as parent time losses and family out-of-pocket costs.
Psychology Inflexibility | 6 weeks
  The Acceptance and Action Questionnaire (AAQ-II) a questionnaire used to measure parent psychological inflexibility or experiential avoidance. The AAQ-II consists of seven items (e.g., "I'm afraid of my feelings," "I worry about not being able to control my worries and feelings") measured on a 1 (never true) to 7 (always true) scale.
Psychology Inflexibility | 4 months
  The Acceptance and Action Questionnaire (AAQ-II) a questionnaire used to measure parent psychological inflexibility or experiential avoidance. The AAQ-II consists of seven items (e.g., "I'm afraid of my feelings," "I worry about not being able to control my worries and feelings") measured on a 1 (never true) to 7 (always true) scale.
Psychology Inflexibility | 12 months
  The Acceptance and Action Questionnaire (AAQ-II) a questionnaire used to measure parent psychological inflexibility or experiential avoidance. The AAQ-II consists of seven items (e.g., "I'm afraid of my feelings," "I worry about not being able to control my worries and feelings") measured on a 1 (never true) to 7 (always true) scale.
Psychology Inflexibility | 18 months
  The Acceptance and Action Questionnaire (AAQ-II) a questionnaire used to measure parent psychological inflexibility or experiential avoidance. The AAQ-II consists of seven items (e.g., "I'm afraid of my feelings," "I worry about not being able to control my worries and feelings") measured on a 1 (never true) to 7 (always true) scale.
Child Development | 18 months
  The Ages and Stages Questionnaire will also be used to assess child development
Parental perception of transition experience | 6 weeks post discharge
  Parental perception of transition experience will be assessed using the Pediatric Transition Experience Measure (PTEM), an 11 item parent-report questionnaire which measures a parent's perception of transition preparation and support from the hospital.

OTHER OUTCOMES:
Health System Outcomes | 12 months
  The investigators will link the patient-reported evaluation of the CCENT model with health administrative data housed at the Institute for Clinical Evaluative Sciences (ICES) for consenting participants. Case-costing methods will be used to determine direct health care costs related to inpatient (emergency department) and outpatient (pharmaceutical and home health care) services.
Social support | Baseline
  The Social Support Questionnaire- Short Form (Sarason et al., 1987) is a 6 item measure of social support. For each of the 6 items, respondents indicate the number of people available to provide support in each of 6 areas and then rate the overall level of satisfaction with the support given in each of the areas. Scores range from 0-54 for number of people available, and satisfaction ranges from 6-36. Higher scores indicate more support.

CONTACTS AND LOCATIONS:
Overall Officials: Julia Orkin, MD, Principal Investigator — The Hospital for Sick Children
Locations (7):
- Canada (7):
  - BC Children's Hospital and BC Women's Hospital & Health Centre, Vancouver, British Columbia
  - Children's Hospital Eastern Ontario, Ottawa, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - The Hospital for Sick Children, Toronto, Ontario
  - Mount Sinai Hospital, Toronto, Ontario
  - McGill University Health Centre/Montreal Children's Hospital, Montreal, Quebec
  - The Ottawa Hospital, Ottawa

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Orkin J, Major N, Esser K, Parmar A, Couture E, Daboval T, Kieran E, Ly L, O'Brien K, Patel H, Synnes A, Robson K, Barreira L, Smith WL, Rizakos S, Willan AR, Yaskina M, Moretti ME, Ungar WJ, Ballantyne M, Church PT, Cohen E. Coached, Coordinated, Enhanced Neonatal Transition (CCENT): protocol for a multicentre pragmatic randomised controlled trial of transition-to-home support for parents of high-risk infants. BMJ Open. 2021 Jul 7;11(7):e046706. doi: 10.1136/bmjopen-2020-046706. PMID 34233983